CLINICAL TRIAL: NCT01363310
Title: A Multi-Centre, Double-Blind, Randomised, Parallel Group, Escitalopram Controlled Phase III-B Study of the Efficacy and Safety of Quetiapine Fumarate Extended Release (Seroquel XR TM) as Monotherapy in the Treatment of Adult Patients With Agitated Major Depressive Disorder
Brief Title: The Quietude Study: Quetiapine Use for Agitated Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination of sponsorship
Sponsor: Physicians Research And Education Network (Other)
Responsible Party: Roger S. McIntyre, MD, FRCPC, Physicians' Research and Education Network
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1443C00037
Record Dates: First submitted 2011-05-20; First posted 2011-06-01 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Depression With Prominent Agitation
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Quetiapine XR (Active Comparator)
  Interventions: Drug: Quetiapine XR
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Quetiapine XR — Dosage form: tablets Day 1-2: 50 mg Day 3-7: 150 mg Day 8-57: either 150 or 300 mg/day (flexible)
  Other Names: Seroquel XR
  Arms: Quetiapine XR
Drug: Escitalopram — Dosage form: capsules Day 1-7: 10 mg Day 8-57: 10 or 20 mg/day (flexible)
  Arms: Escitalopram

SUMMARY:
Most individuals with major depressive disorder manifest clinically significant agitation. Concurrent agitation in a depressed individual is associated with an intensification of mood symptoms, decreased probability of recovery, increased recurrence risk, suicidality, and increased medical-service utilization. The occurrence of anxiety/agitation phenomenology in the depressed patient often invites the need for augmentation strategies (e.g. atypical antipsychotics, benzodiazepines, etc.) and complicated polypharmacy regimens. Moreover, individuals with major depressive disorder often report worsening of symptom severity, irritability, hostility, dysphoria, and significant subjective distress (This response pattern is similar to individuals with bipolar disorder).

Results from large research studies provide evidence indicating that quetiapine is capable of offering clinically significant multidimensional symptom relief in bipolar depression. Moreover, results from several trials in major depressive disorder and generalized anxiety disorder have established the efficacy of quetiapine therapy for unipolar depression and anxiety syndromes. So far, no atypical antipsychotic agent has been evaluated specifically for the treatment of agitated depression.

In this study, it is hypothesized that persons with major depressive disorder and prominent agitation (i.e. agitated depression) will exhibit a more favourable response and tolerability profile to quetiapine XR when compared to escitalopram.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 to 65
* Outpatient at enrolment
* A diagnosis of major depressive disorder
* Baseline HAMD-17 score > 20 and HAMD Item1 score > 2 both at enrolment and baseline
* Significant agitation
* CGI-S score > 4 at screening and baseline
* Negative serum pregnancy test at enrolment and use of a reliable method of birth control during the study
* Able to understand and comply with the requirements of the study
* Able and willing to give meaningful informed written consent

Exclusion Criteria:

* Another Axis I diagnosis of primary focus within 6 months of enrolment
* Axis II disorder causing impact on current diagnosis
* Current depressive episode <4 weeks, or >12 months
* Substance or alcohol abuse or dependency as defined by DSM IV within 6 months of enrolment
* Any pervasive developmental disorder or dementing disorder
* Treatment with other antipsychotics, mood stabilizer or other psychoactive drugs less than 7 days prior to randomization
* Treatment with fluoxetine less than 28 days prior to baseline
* Treatment with MAO inhibitors, anxiolytic drugs in excess of 2 mg lorazepam equivalents/day.
* Insufficient response to more than two antidepressants during the index episode prior to study involvement
* Known lack of antidepressant response to quetiapine at a dose of at least 50 mg/day x 4 weeks
* Known lack of antidepressant response to escitalopram at a dose of at least 10 mg/day
* Known intolerance or hypersensitivity to quetiapine or escitalopram
* Treatment with Electroconvulsive therapy within 90 days prior to baseline
* Use of Potent P450 3A4 inhibitors or inducers within 14 days of baseline
* AST & ALT ≥ 3X ULN
* TSH ≥ 10% ULN
* Unstable medical condition
* Medical condition the would affect absorption, distribution, metabolism or excretion of study treatment
* Significant ECG abnormalities
* Pregnancy or lactation
* Patients with increased suicidal risks, HAM-D item 3 ≥3 or have made a suicide attempt within the past 6 months.
* Patients who, in the investigators opinion, will require psychotherapy (other than supportive psychotherapy) during the study period, unless psychotherapy has been ongoing for a minimum of 3 months prior to randomisation
* A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:
* Unstable DM defined as enrolment glycosylated haemoglobin (HbA1c) >8.5%.
* Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
* Not under physician care for DM.
* Physician responsible for patient's DM care has not indicated that patient's DM is controlled.
* Physician responsible for patient's DM care has not approved patient's participation in the study
* Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 weeks.
* Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study
* Clinically significant deviation from the reference range in clinical laboratory test results
* An absolute neutrophil count (ANC) of 1.5 x 109 per liter
* Those who are involved in the planning and/or conduct of the study cannot be enrolled as subjects
* Previous enrolment or randomization in the present study
* Participation in another medication trial within 4 weeks prior to enrolment into the study herein

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to endpoint in the Hamilton Depression Rating Scale 17-Item (HAMD-17) total score | Day 1, Day 57
  A tool to assess the range of symptoms of depression

SECONDARY OUTCOMES:
Change in anxiety factor score on the Hamilton Depression Rating Scale 17-item (HAMD-17) from baseline to endpoint | Day 1, Day 57
  A tool to assess the range of symptoms of depression
Change from baseline to endpoint in Hamilton Anxiety Rating Scale (HAMA) total score | Day 1, Day 57
  A tool to measure severity of symptoms of anxiety
Change in Clinical Global Impression score from baseline to endpoint | Screening Visit, Day 1, Day 8, Day 15, Day 29, Day 43, Day 57
  A tool to assess illness severity, improvement and response to treatment
Change from baseline to endpoint in Sheehan Disability Scale (SDS) sub-scales and total score | Day 1, Day 57
  A tool to assess functional impairment
Change in Hamilton Depression Rating Scale 17-item (HAMD-17) sleep disturbance factor score on the from baseline to endpoint | Day 1, Day 57
  A tool to assess the range of symptoms of depression
Change in Hamilton Anxiety Rating Scale (HAMA) somatic and psychic anxiety factor scores from baseline to endpoint | Day 1, Day 57
  A tool to measure severity of symptoms of anxiety
Change from baseline in the Sex Functioning Questionnaire (Sex FX) | Day 1, Day 57
  A tool to assess sexual functioning
Change in blood pressure and heart rate from baseline to end of treatment | Day 1, Day 57
Change in weight, BMI, waist circumference from baseline to end of treatment | Day 1, Day 57
Change in findings from physical examination from baseline to end of treatment | Screening, Day 57
Tabulation of spontaneous adverse events | Day 1, Day 57
Tabulation of clinical haematology and chemistry results | Screening, Day 57
Incidence of premature study withdrawal due to inadequate control of depressive symptoms
Proportion of patients with HAM-D Item 3 score > 2 at any time after randomization or adverse events of suicidality/suicidal ideation/suicide attempts/suicide completion | Day 1, Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, MD, FRCPC, Study Director — Physicians Research And Education Network
Locations (11):
- Canada (11):
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - Aptekar Medicine Professional Corporation, Brampton, Ontario
  - Chatham-Kent Health Alliance, Chatham, Ontario
  - Fort Erie Group Family Practice, Fort Erie, Ontario
  - Brady Clinic, Greater Sudbury, Ontario
  - Georgina Family Medical Centre, Keswick, Ontario
  - Richmond Oxford Walk-In Clinic, London, Ontario
  - Gerald Rockman Medicine Professional Corporation, Scarborough Village, Ontario
  - Bloor-Park Medical Centre, Toronto, Ontario
  - Primary Care Lung, Toronto, Ontario
  - Manna Research, Toronto, Ontario